CLINICAL TRIAL: NCT05645471
Title: Comparative Effectiveness of Together After Cancer Among Breast Cancer Survivors and Their Intimate Partners
Brief Title: Together After Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); University of Miami Sylvester Comprehensive Cancer Center (Other); AdventHealth (Other); University of Central Florida (Other)
Responsible Party: Principal Investigator, Dinorah Martinez Tyson, PhD, MPH, MA, Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 004181; AD-2020C3-21171 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2022-10-12; First posted 2022-12-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Quality of Life; Communication
Keywords: Breast Cancer, Latino, Couples,
MeSH Terms: conditions — Breast Neoplasms; Communication

STUDY DESIGN:
Intervention Model Description: The study aims to test the impact of the adapted Together After Cancer intervention using a cluster randomized controlled trial (cRCT), with individuals nested within couples and randomization occurring at the couple level to see if it is more effective than usual care (UC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Together After Cancer Intervention (Experimental): Couples randomized into the intervention will participate in the program which is approximately 8-10 hours of web-based online content to be delivered over the course of 5-8 weeks. The online program can be done on a smartphone, tablet, or computer. In this program, partners complete the majority of the program on their own (to make it more flexible) and come together for 2-3 key conversations with their partner. In addition to the online content, couples will receive up to 100 minutes of scheduled research check-in/coaching calls from a research assistant to check-in. These coach calls will occur via a video chat via Zoom or, if not possible given a couple's technology limitations, over the phone. The coach calls serve several purposes: a) helping couples stay accountable to staying on the recommended schedule of activity completion; b) addressing any technical or program questions the couple has; and c) collecting research data as couples move through the program.
  Interventions: Behavioral: Together After Cancer
- Usual Care (No Intervention): Participants randomized into UC, will consist of primary referral sources for breast cancer survivorship. At AdventHealth, Moffitt, and Sylvester Cancer centers, usual care consists of screening items assessing relationship/intimacy issues as a practical need. If these items are endorsed, referrals are provided to supportive oncology. At Sylvester, the Cancer Support Services offers caregiver support groups, "mental well-being" services (i.e., individual therapy), and an online support community for patients, caregivers, and survivors. At Moffitt, Support Services offers psychotherapy, support groups for patients, support groups for family/caregivers of cancer patients, and a program to help patients talk with their children about their diagnosis. At AdventHealth, patients are offered referrals to social services and psychoeducational programs like HEAL. However, none of the sites have services designed to focus on issues specific to patients' romantic relationships.

INTERVENTIONS:
Behavioral: Together After Cancer — This is an online couples intervention for Latina breast cancer survivors and their intimate partners.
  Arms: Together After Cancer Intervention

SUMMARY:
To evaluate the impact of an adapted online, self-help relationship intervention (supplemented with brief coach calls) for survivors of breast cancer and their partners. Couples will be randomized to receive either the online intervention (Together after Cancer) or usual care (UC) and assessed at baseline, end of the program, and 3 months after randomization.

DETAILED DESCRIPTION:
As the fastest-growing and largest ethnic minority group, projections indicate that 128 million Latinos will reside in the United States by 2050; with one in three Latinos receiving a diagnosis of cancer during his/her lifetime. Latino cancer survivors have a lower quality of life, experience distress due to strained spousal and family relationships, have poorer physical health, and have more depression, pain, and fatigue when compared to non-Latinos. In addition, emotional and mental well-being between Latino survivors and their partners is related, with partners also experiencing increased distress and physical symptoms. Research has shown that couples-based psychosocial programs improve the quality of life and emotional and physical health of cancer survivors and their partners. Yet, much of the in this area has focused on non-Hispanic Whites. Features of Latino culture may influence and interact with social, psychosocial, health care, and clinical factors that influence cancer-related outcomes. Our goal is to add to this literature and develop a program for Latina breast cancer survivors and their partners that is culturally meaningful and relevant and responds to their needs and concerns.

Specifically, investigators plan to culturally adapt a widely-available and effective online couple intervention, OurRelationship (ORI), for Latina breast cancer survivors and their intimate partners. The online OR program - which can be done on a smartphone, tablet, or computer - was developed to serve as an online tool to help couples solve a specific relationship problem they selected. Investigators will adapt the OR program to be useful for Latina breast cancer survivors and their intimate partners using feedback from focus groups with patients, community partners, and research advisors. Once investigators have completed our adaptation, the plan to test the impact of the adapted program, Together after Cancer, using a type of study called a randomized controlled trial where participants will be randomly allocated to either receive the culturally adapted intervention or usual care. Investigators are interested in learning if couples in the group that are assigned to the intervention program report changes in their relationship functioning, psychological functioning (depression, anxiety, and perceived stress), and cancer-related quality of life (pain, fatigue, body image, and quality of life) compared to couples who are assigned to the UC group.

Through this comparative study, investigators expect to establish effective strategies that can be implemented in clinic and community settings to improve psychological functioning, relationship functioning, and quality of life. Investigators are enthusiastic about the potential for the intervention program to easily reach cancer Latina survivors around the nation, due to the online format and ease of access from any location. Throughout the project, investigators will continue to engage our local partners to ensure that the study procedures and outcomes are meaningful to all stakeholders.

Investigators are using patient-centered approaches to offer a culturally relevant web-based program that cancer survivors and their partners can access from the comfort of their homes.

ELIGIBILITY:
Inclusion Criteria for Latina Breast Cancer Survivors:

* Be 18 years of age and older
* Self-identify as Latina/Hispanic
* Spanish or English speaker
* Primary diagnosis of breast cancer in the last ten years
* Completed initial treatment
* Be married or in a committed relationship of six months duration or longer
* Willingness to be randomized and followed for approximately 5 months
* Access to the internet or a smartphone, tablet, or computer

Inclusion criteria for Intimate Partners:

* Be 18 years of age or older
* Be married or in a committed relationship of six months duration or longer with a Latina Breast Cancer Survivor diagnosed who was diagnosed with breast cancer in the last ten years
* Willingness to be randomized and followed for approximately 5 months
* Access to the internet or a smartphone, tablet, or computer

Couples will be eligible to participate if they also meet the following:

* Meet the inclusion criteria listed above for Latina Breast Cancer Survivors and Intimate Partners
* Both partners are willing to participate in the study
* Additionally, to be eligible, the Latina Breast Cancer Survivors must reside in Florida

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the changes in the quality of life of the breast cancer survivor across the pre to post to follow-up measurement time points. | Baseline, 2 and 5 month
  The FACT-B is a 37-item instrument designed to measure five domains of HRQOL in breast cancer patients which focuses on physical, social, emotional, functional well-being as well as a breast-cancer subscale. Each question is rated on a four-point scale from 0=Not at all to 4=Very Much. The scale has an internal consistency of an α=.90, with subscale alpha coefficients ranging from .63 to .86.
Evaluate the changes in the satisfaction of the relationship between couples who are married across the pre to post to follow-up measurement time points. | Baseline, 2 and 5 month
  The Couples Satisfaction Index (CSI) is a 32- item instrument assess one's satisfaction in a relationship which assess the presence of problems between individuals and the intensity of such problems. Each question is rated on a six-point scale from 0=Extremely Unhappy to 6=Perfect. The scale as an internal consistency α=0.92.

SECONDARY OUTCOMES:
Evaluate the changes in the cancer-related body image of the breast cancer survivor across the pre to post to follow-up measurement time points. | Baseline, 2 and 5 month
  The Body Image Scale is a 10-item measure developed to measure cognitive, affective, and evaluative variables of an individual's concept of body image and reflects relatively time-stable physical aspects, rather than current physical conditions. Each question is rated on a four-point scale from 1=Not at all to 4=Very much. The scale has an internal consistency is α=.90.
Evaluate the changes in cancer-related fatigue of the breast cancer across the pre to post to follow-up measurement time points. | Baseline, 2 and 5 month
  The Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue is a 7-item scale that assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Each question is rated on a four-point scale from 1=Not at all to 4=Very much. The scale has an internal consistency is α=0.79.
Evaluate changes in the quality of life among the intimate partner across the pre to post to follow-up measurement time points. | Baseline, 2 and 5 month
  The Functional Assessment of Cancer Therapy-General Pop. (FACT-GP) a shortened, 21-item that assess the perceived levels of health-related quality of life in the partner. Each question is rated on a five-point scale from 0=Not at all to 4=Very much. The scale has an internal consistency is α=0.89.
Evaluate changes in emotional distress-depression among breast cancer survivor and their intimate partner across the pre to post to follow-up measurement time points. | Baseline, 2, 5 month
  The PROMIS: Emotional Distress-Depression is an 8-item survey related to depressed mood in the past 7 days. Each question is rated on a five-point scale from 1=Never to 5=Always. The internal consistency is α=0.97.
Evaluate changes in emotional distress-anxiety among breast cancer survivors and their intimate partner across the pre to post to follow-up measurement time points. | Baseline, 2, 5 month
  The PROMIS: Emotional Distress - Anxiety is a 6-item survey that assess self-reported fear, anxious misery, hyperarousal and somatic symptoms related to arousal. Each question is rated on a five-point scale from 1=Never to 5=Always. The internal consistency is α=0.96.
Evaluate changes in stress among breast cancer survivors and their intimate partner across the pre to post to follow-up measurement time points. | Baseline, 2, 5 month
  The Perceived Stress Scale (PSS) is a 10-item that measures the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. Each question is rated on a five-point scale from 0=never to 4 very often. The internal consistency is α=0.74.
Evaluate changes in feeling cared and valued as a person among breast cancer survivors and their intimate partner across the pre to post to follow-up measurement time points. | Baseline, 2, 5 month
  The PROMIS: Emotional Support is a 4-item that assess perceived feelings of being cared and valued as a person; having confidant relationships. Each question is rated on a five-point scale from 1=Never to 5=Always. The internal consistency is α=0.98.
Evaluate changes in supportive communication among breast cancer survivors and their intimate partner across the pre to post to follow-up measurement time points. | Baseline, 2, 5 month
  The Dyadic Coping Inventory is a 37-item instrument designed to measure perceived communication and dyadic coping (supportive, delegated, negative, and joint) that occurs in close relationships when one or both partners are stressed. The internal consistency is α=0.86.
Evaluate changes in negative communication between the breast cancer survivor and their intimate partner across the pre to post to follow-up measurement time points. | Baseline, 2, 5 month
  The Conflictual Communication Index is a 7-item measure developed to assess negative communication. Participants were asked to report how often communication conflict occurred during the past month on a Likert-type scale from 1=Never to 4= Often. The internal consistency is α=0.89.
Evaluate changes in intimacy between the breast cancer survivor and their intimate partner across the pre to post to follow-up measurement time points. | Baseline, 2, 5 month
  The Personal Assessment of Intimacy in Relationships (PAIR) is a 6-item measure of that assesses comfort, intimacy, and satisfaction with sexual relationship of a couple. Each question is rated on a five-point scale from 1=Very rarely to 5=Very often. The internal consistency is α=0.86.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sylvester Comprehensive Cancer Center and University of Miami, Miami, Florida
  - AdventHealth, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No